CLINICAL TRIAL: NCT05647226
Title: Exploring the Use of Digital Therapeutics Alongside a Remote Intensive Lifestyle Programme on Inducing Weight Loss and Diabetes Remission in Patients With Type 2 Diabetes Versus Standard of Care (DIGEST)
Brief Title: Digital Diabetes Remission Trial
Acronym: DIGEST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Habitual Health Ltd (Industry)
Collaborators: Lindus Health (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 312269
Record Dates: First submitted 2022-11-30; First posted 2022-12-12 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: A multicentre, open-label, parallel design, randomised controlled trial.
Who Masked: Outcomes Assessor
Masking Description: Due to the nature of the lifestyle programme, participants, clinicians and data collectors will not be able to be masked, however allocation will be concealed from the statistician in charge of performing the analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention arm (Experimental): Intervention participants will be given an initial 12-week low energy-diet (LED) and will have continual use of an intensive behaviour education programme delivered through an app.
  Interventions: Combination Product: Digital therapeutic and intensive lifestyle programme
- Standard of care arm (Other): All participants in the control arm will receive standard care provided by the National Health Service.
  Interventions: Other: Standard of care

INTERVENTIONS:
Combination Product: Digital therapeutic and intensive lifestyle programme — Initial 12-week LED and behaviour education app.
  Arms: Intervention arm
Other: Standard of care — Standard of care.
  Arms: Standard of care arm

SUMMARY:
This is a multicentre, open-label Randomised Controlled Trial run in the United Kingdom. The main aims are to assess whether the Habitual Remission Programme (digital therapeutics + 12-week 800kcal/day low-energy diet, delivered remotely) is more likely to lead to weight loss and remission in adults with type 2 diabetes, when compared to standard of care.

DETAILED DESCRIPTION:
Participants will be randomly allocated to the Habitual Programme or standard care as delivered by the National Health Service (NHS). They will take a home blood test for HbA1c at baseline, 3 months and 6 months, and complete online fortnightly surveys to record their weight, waist circumference, blood pressure, side-effects and any changes in medication, for 6 months. These measurements will be taken at 6 months and 12 months after finishing the intervention for those allocated to the intervention.

Participants will be recruited from General Practitioner (GP) surgeries in England, managed by Lindus Health. Research Nurses at Lindus Health will complete screening and informed consent procedures.

ELIGIBILITY:
Inclusion Criteria:

* Able and willing to give consent for the study prior to participation
* Be aged between 18-75 years, with type 2 Diabetes Mellitus of duration <6years.
* Has access to a smartphone or computer
* Has a Body Mass Index (BMI) of ≥28 kg/m2
* HbA1C between 86 mmol/mol (10%) ≥ 48mmol/mol (6.5%), within the previous 12-months

Exclusion Criteria

* Is currently using Insulin
* Weight of change >5% in the past 3-months
* Has a history of are known to be suffering with alcohol/substance abuse
* Has cancer or is knowingly under investigation for cancer
* Has had a myocardial infarction within the previous 6-months
* Has severe or unstable heart failure e.g., New York Heart Association (NYHA) grade IV
* Has porphyria
* Has learning difficulties
* Is currently on treatment with anti-obesity drugs
* Has had bariatric surgery
* Has been diagnosed with an eating disorder or purging
* Is pregnant or less than 4-months postpartum or considering pregnancy in the next 2-years
* Is currently breastfeeding
* Has required hospitalisation for depression or taking antipsychotic drug
* Has a history of illnesses that could interfere with the interpretation of the study (e.g. HIV, Cushing syndrome, chronic kidney disease, chronic liver disease, hyperthyroidism, hereditary fructose intolerance, depression or antipsychotic drug use within the past 2 years)
* Currently talking Glucagon-like peptide-1 receptor agonists (GLP-1 RAs)
* Has pancreatitis
* Currently taking part in a Clinical Trial of an Investigative Medicinal Product (CTIMP) trial for antidiabetic medication
* Abnormal diabetic foot review (QOF codes for diabetic foot at moderate risk, at high risk, at increased risk, ulcerated).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2022-01-09 (Actual); Primary Completion 2024-07-30 (Actual); Study Completion 2024-07-30 (Actual)

PRIMARY OUTCOMES:
Weight loss of ≥15kg | 6-months
  Number of participants that achieved ≥15kg
HbA1C <6.5% (48mmol/mol) | 6-months
  Number of participants who have achieved HbA1C <6.5% (48mmol/mol) after at least 2-months of all glucose-lowering medication.

SECONDARY OUTCOMES:
Glycaemic Control | 3-months- 6-months
  Changes in HbA1C from baseline to mid and endpoints.
Weight control | 3-months- 6-months
  Changes in weight from baseline to mid and endpoints.
Systolic blood pressure (SBP) | 3-months- 6-months
  Changes in SBP from baseline to mid and endpoints.
Diastolic blood pressure (DBP) | 3-months- 6-months
  Changes in DBP from baseline to mid and endpoints.
Medication use | Baseline, 3-months and 6-months
  Medication use reported by the participant.
Weight loss ≥10kg | 6-months
  Number of participants that achieved ≥10kg
Safety of Intervention | Baseline- 6-months
  Monitoring the number of Adverse Events (AEs), Severe Adverse Events (SAEs) and (S)AE's that constitute Major Adverse Cardiovascular Events and Major Adverse Diabetes Events
HbA1C <6.5% (48mmol/mol) | 12-months (6-months after completing the trial).
  Number of participants with an HbA1C <6.5% (48mmol/mol) after a 6-month follow up

CONTACTS AND LOCATIONS:
Overall Officials: Carol Le Roux, Professor, Principal Investigator — Principal Investigator
Locations (1):
- Lindus Health Ltd, London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Data will be entered into a validated Electronic Data Capture (EDC) platform. Direct access to the EDC platform will be granted to authorised representatives from the Sponsor, Lindus Health and the regulatory authorities to allow trial-related monitoring, audits and inspections.

REFERENCES:
- [Background] Lean ME, Leslie WS, Barnes AC, Brosnahan N, Thom G, McCombie L, Peters C, Zhyzhneuskaya S, Al-Mrabeh A, Hollingsworth KG, Rodrigues AM, Rehackova L, Adamson AJ, Sniehotta FF, Mathers JC, Ross HM, McIlvenna Y, Stefanetti R, Trenell M, Welsh P, Kean S, Ford I, McConnachie A, Sattar N, Taylor R. Primary care-led weight management for remission of type 2 diabetes (DiRECT): an open-label, cluster-randomised trial. Lancet. 2018 Feb 10;391(10120):541-551. doi: 10.1016/S0140-6736(17)33102-1. Epub 2017 Dec 5. PMID 29221645
- [Background] Lean MEJ, Leslie WS, Barnes AC, Brosnahan N, Thom G, McCombie L, Peters C, Zhyzhneuskaya S, Al-Mrabeh A, Hollingsworth KG, Rodrigues AM, Rehackova L, Adamson AJ, Sniehotta FF, Mathers JC, Ross HM, McIlvenna Y, Welsh P, Kean S, Ford I, McConnachie A, Messow CM, Sattar N, Taylor R. Durability of a primary care-led weight-management intervention for remission of type 2 diabetes: 2-year results of the DiRECT open-label, cluster-randomised trial. Lancet Diabetes Endocrinol. 2019 May;7(5):344-355. doi: 10.1016/S2213-8587(19)30068-3. Epub 2019 Mar 6. PMID 30852132
- See also: Habitual Health Ltd (Sponsor) — https://www.tryhabitual.com/